CLINICAL TRIAL: NCT07119866
Title: The Role of Oxygen Reserve Index (ORi) Monitoring in Optimizing Apneic Ventilation for Laparoscopic Cholecystectomy
Brief Title: The Role of Oxygen Reserve Index (ORi) in Apneic Ventilation
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayça Özcan, Prof., Ankara City Hospital Bilkent
Other Study IDs: Oxygen Reserve Index
Record Dates: First submitted 2025-07-21; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Oxygen Reserve Index; Apnea; Ventilation; Body Mass Index
MeSH Terms: conditions — Apnea; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ORI>0.24: Patients, aged between 18 and 60 years, classified as ASA physical status I-II,and with a Mallampati score <2, were enrolled.On the day of surgery, following identity verification and confirmation of the surgical site, patients were positioned on a warmed operating table.Standard monitoring was applied, including ECG, SBP and DBP, SpO₂, and the ORI.Preoxygenation was achieved by administering 100% oxygen via 8 deep breaths over 60 seconds.When the ORI value reached 0.4, intravenous anesthesia induction was initiated using propofol 2 mg/kg, fentanyl 2 mcg/kg, and rocuronium 0.6mg/kg.During muscle relaxation, patients were not ventilated via mask.The ORI value at the time of induction and at the 2nd minute post-induction was recorded.If the ORI dropped below 0.24 before the 2-minute mark, mask ventilation was initiated, and the time of intervention was noted.Endotracheal intubation was then performed using a standard,atraumatic technique after achieving adequate muscle relaxation.
  Interventions: Other: OXYGEN RESERVE INDEX
- ORI<0.24: Patients, aged between 18 and 60 years, classified as ASA physical status I-II,and with a Mallampati score <2, were enrolled.On the day of surgery, following identity verification and confirmation of the surgical site, patients were positioned on a warmed operating table.Standard monitoring was applied, including ECG, SBP and DBP, SpO₂, and the ORI.Preoxygenation was achieved by administering 100% oxygen via 8 deep breaths over 60 seconds.When the ORI value reached 0.4, intravenous anesthesia induction was initiated using propofol 2 mg/kg, fentanyl 2 mcg/kg, and rocuronium 0.6mg/kg.During muscle relaxation, patients were not ventilated via mask.The ORI value at the time of induction and at the 2nd minute post-induction was recorded.If the ORI dropped below 0.24 before the 2-minute mark, mask ventilation was initiated, and the time of intervention was noted.Endotracheal intubation was then performed using a standard,atraumatic technique after achieving adequate muscle relaxation.
  Interventions: Other: OXYGEN RESERVE INDEX

INTERVENTIONS:
Other: OXYGEN RESERVE INDEX — Noted for each patient.

SUMMARY:
Background: The Oxygen Reserve Index (ORI) is a non-invasive parameter utilizing multi-wavelength pulse co-oximetry. ORI can provide early warnings of deteriorating oxygenation before changes are reflected in SpO₂ levels. This study aimed to investigate the feasibility of non-ventilated intubation in patients undergoing cholecystectomy as a means to achieve safe intubation without nasogastric tube placement, with reduced trauma and cost, and improved time efficiency.

DETAILED DESCRIPTION:
Obesity is a complex and chronic disease that significantly impacts respiratory physiology. It leads to increased work of breathing and reduced compliance of the chest wall. In morbidly obese individuals, there is a marked reduction in total lung capacity, vital capacity, forced expiratory volume in one second (FEV1), and forced vital capacity (FVC). Additionally, due to their elevated metabolic demands, these patients exhibit higher oxygen consumption rates.

The Oxygen Reserve Index (ORi) (Masimo Corp., Irvine, CA, USA) is an advanced, continuous, and non-invasive parameter that provides a relative indication of arterial partial pressure of oxygen (PaO₂).

ORI monitoring can be particularly beneficial in patients at risk for inadequate preoxygenation, those with difficult mask ventilation, hypoxemic patients with aspiration risk, rapid sequence induction scenarios, obese individuals, ICU intubations, and invasive ventilation cases. It has also been shown to provide early warnings of desaturation in select patient groups, contributing to improved patient safety.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* ASA 1-2
* Mallampati score <2
* Scheduled for elective laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* <18 and >60 years
* ASA 3-4
* Initial ORI value below 0.24

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 60 patients between the ages of 18-60 years, ASA 1-2, scheduled for elective laparoscopic cholecystectomy under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-07 (Estimated); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
TIME FOR ORI TO FALL BELOW 0.24 | WITHIN 10 MINUTES BEFORE INTUBATION
  TIME THE PATIENT STARTED TO WEAR A MASKS.

SECONDARY OUTCOMES:
INITIAL ORI VALUE | WITHIN 10 MINUTES BEFORE INTUBATION
  Noted for each patient.
ORI VALUE AT 2 MINUTES | WITHIN 10 MINUTES BEFORE INTUBATION
  Noted for each patient.
AGE | WITHIN 10 MINUTES BEFORE INTUBATION
  Noted for each patient.
American Society of Anesthesiologists (ASA) Score | WITHIN 10 MINUTES BEFORE INTUBATION
  Noted for each patient.
SEX | WITHIN 10 MINUTES BEFORE INTUBATION
  Noted for each patient.
BMI | WITHIN 10 MINUTES BEFORE INTUBATION
  Noted for each patient.
PRESENCE OF A NASOGASTRIC TUBE | 10 MINUTES BEFORE EXTUBATION
  Noted for each patient.
Surgeon satisfaction | 10 MINUTES BEFORE EXTUBATION
  Noted for each patient. Surgeon satisfaction according to ng usage status.
PRESENCE OF LARYNGOSPASM | 10 MINUTES BEFORE EXTUBATION
  Noted for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, çankaya, Turkey (Türkiye)